CLINICAL TRIAL: NCT03035110
Title: A Feasibility Study to Evaluate Self-Harm Group in Inpatient Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Essex (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 205350
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Self-Injurious Behavior
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dialectical Behavioural Therapy (DBT) skills group (Experimental): Four group sessions, based on DBT, over two weeks, with a group of four to eight participants in attendance located on the hospital ward where the participant is a patient.
  Interventions: Behavioral: Dialectical Behavioural Therapy (DBT) based skills groups

INTERVENTIONS:
Behavioral: Dialectical Behavioural Therapy (DBT) based skills groups — Dialectical Behavioural Therapy (DBT) involves skills that help people manage their emotions and tolerate distress. This therapy is found effective in reducing self-harm behaviour for outpatients with Borderline Personality Disorder.

SUMMARY:
The current research is being undertaken as part of a professional doctorate in clinical psychology, which aims to evaluate the feasibility of a group programme to address self-harm within 23 days, to provide evidence for a controlled trial. The intervention will include four group sessions conducted over 2 weeks, based on Dialectical Behavioural Therapy. Specifically the aims are to determine 1) means and a standard deviation for two pre and post treatment outcome measures in order to estimate sample size for the main study, 2) the need for an inpatient intervention for self-harm measured by number of participants eligible and accepting of the treatment, 3) retention of participants for 4 groups given the predicted short stays of patients on wards, and 4) the acceptability of the research process for this client group through feedback.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be screened by their allocated clinician and included if they are aged between 18-65
* admitted to hospital
* have a history of or engaged in at least one episode of self-harm, iv) have capacity to understand the information sheet.

Exclusion Criteria:

* Participants will be screened by clinicians and they will exclude people if i) they are Non-English speakers (due to translation costs)
* they lack the capacity to give informed consent (assessed by their key clinician)
* their symptoms prevent them from concentrating for an hour at a time (i.e. severe thought disorder), and therefore not benefiting from the group (assessed by their key clinician)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
The Inventory of Statements About Self-Injury (ISAS) | 23 days
  ISAS is a self-report measure designed to assess the function and frequency of deliberate self-harm. It will be administered pre- and post-intervention.
The Distress Tolerance Scale (DTS) | 23 days
  The DTS consists of 15 items, which measure a person's appraisal of their emotional distress, their ability to tolerate this distress and any regulation efforts to alleviate it. It will be administered pre- and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Goodmayes Hospital, Ilford, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No